CLINICAL TRIAL: NCT02783027
Title: Real-time Fatigue Mitigation With Air-medical Personnel: The SleepTrackTXT2 Randomized Trial
Brief Title: The SleepTrackTXT2 Randomized Trial With Air-medical Personnel
Acronym: SleepTrack2
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pittsburgh (Other)
Responsible Party: Principal Investigator, Daniel Patterson, PhD, NRP, Assistant Professor, University of Pittsburgh
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: PRO16030345
Record Dates: First submitted 2016-05-23; First posted 2016-05-26 (Estimated); Results first posted 2019-12-26 (Actual); Last update posted 2019-12-26 (Actual); Status verified 2019-12

CONDITIONS: Poor Quality Sleep; Fatigue
MeSH Terms: conditions — Fatigue

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- SleepTrackTXT2 (Experimental): Participants will receive text-message based assessment during shift work (intra-shift) and between shifts (inter-shift). Participants in the experimental group that report high levels of fatigue, sleepiness, or difficulty with concentration during shift work (intra-shift) will receive tailored text-messages promoting adoption of behaviors that can improve alertness. Participants will also receive a summary of their sleep debt once a week and suggestions for paying back sleep debt. Participants will also have access to a graphic summary of their sleep hours over previous 30-days.
  Interventions: Behavioral: SleepTrackTXT2
- Text-Message Assessments Only (No Intervention): Participants in the non-intervention group/arm will receive text-message based assessment during shift work (intra-shift) and between shifts (inter-shift). The inter-shift assessments will query the participant about his/her sleep hours, fatigue, sleepiness, and difficulty with concentration. No intervention messages sent to this group/arm.

INTERVENTIONS:
Behavioral: SleepTrackTXT2 — Participants that report high levels of fatigue, sleepiness, or difficulty with concentration during shift work (intra-shift) will receive tailored text-messages promoting adoption of behaviors that can improve alertness during shift work. Participants will also receive a summary of their sleep debt once a week and suggestions for paying back sleep debt. Participants will also have access to a graphic summary of their sleep hours over previous 30-days.
  Arms: SleepTrackTXT2

SUMMARY:
The overarching goal of this proposal is to address the MedEvac foundation priority of educational techniques and technologies and improve Helicopter Emergency Medical Services (HEMS) safety by determining if overall sleep quality and intra-shift fatigue of HEMS clinicians can be improved with real-time assessment and intervention.

Aim 1: To determine the short-term impact of an enhanced SleepTrackTXT intervention on HEMS clinician fatigue reported in real-time during and at the end of shift work.

Aim 2: To determine the long-term impact of the SleepTrackTXT intervention on sleep quality and sleep health indicators including hours of sleep and recovery between shift work.

DETAILED DESCRIPTION:
The investigators will examine short term impact by examining self-reported fatigue captured at the start, during, and end of scheduled shifts.

The investigators will determine longer-term impact on sleep quality by comparing scores on the Pittsburgh Sleep Quality Index (PSQI) taken at baseline and then again at 4 months.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age and older
* working clinically at a study site
* currently working in shifts
* has a smart phone and
* willing to take part in a research study that requires the sending and receiving of multiple text messages daily over 4-months

Exclusion Criteria:

* does not meet inclusion criteria

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 83 (Actual)
Dates: Start 2016-06 (Actual); Primary Completion 2017-08 (Actual); Study Completion 2017-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Patterson, PhD, Principal Investigator — University of Pittsburgh
Locations (1):
- University of Pittsburgh Medical Center / STAT MedEvac, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No
Do not plan to share data unless required by the MedEvac Foundation

REFERENCES:
- [Background] Patterson PD, Moore CG, Guyette FX, Doman JM, Sequeira D, Werman HA, Swanson D, Hostler D, Lynch J, Russo L, Hines L, Swecker K, Runyon MS, Buysse DJ. Fatigue mitigation with SleepTrackTXT2 in air medical emergency care systems: study protocol for a randomized controlled trial. Trials. 2017 Jun 5;18(1):254. doi: 10.1186/s13063-017-1999-z. PMID 28583143
- [Result] Patterson PD, Moore CG, Guyette FX, Doman JM, Weaver MD, Sequeira DJ, Werman HA, Swanson D, Hostler D, Lynch J, Russo L, Hines L, Swecker K, Kroemer AJ, Runyon MS, Buysse DJ. Real-Time Fatigue Mitigation with Air-Medical Personnel: The SleepTrackTXT2 Randomized Trial. Prehosp Emerg Care. 2019 Jul-Aug;23(4):465-478. doi: 10.1080/10903127.2018.1532476. Epub 2018 Oct 29. PMID 30285519

RESULTS

PARTICIPANT FLOW:
Groups:
- SleepTrackTXT2: Participants receive text-message assessment during shift work (intra-shift) and between shifts (inter-shift). Participants in the experimental group that report high levels of fatigue, sleepiness, or difficulty with concentration during shift work (intra-shift) will receive tailored text-messages promoting adoption of behaviors that can improve alertness. Participants will also receive a summary of their sleep debt once a week and suggestions for paying back sleep debt. Participants will also have access to a graphic summary of their sleep hours over previous 30-days.
Period: Overall Study
Arm/Group | SleepTrackTXT2 | Text-Message Assessments Only
Started | 39 | 44
Completed | 16 | 27
Not Completed | 23 | 17

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | SleepTrackTXT2 | Text-Message Assessments Only | Total
Number analyzed (Participants) | 39 | 44 | 83
Age, Continuous [Mean (Standard Deviation); unit: years] — Population: 2 participants in each group did not complete the age information
  years
    number analyzed (Participants) | 37 | 42 | 79
    (all) | 40.9 (9.5) | 41.8 (9.8) | 41.4 (9.7)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: 1 participant in the intervention group and 2 in the control did not complete sex information
  Participants
    number analyzed (Participants) | 38 | 42 | 80
    Female | 19 | 15 | 34
    Male | 19 | 27 | 46
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Most Common Shift Length [Count of Participants; unit: Participants] — Population: 1 participant in each group did not complete the shift length question on the baseline assessment.
  Participants
    number analyzed (Participants) | 38 | 43 | 81
    24 Hours | 18 | 21 | 39
    12 Hours | 18 | 22 | 40
    Other | 2 | 0 | 2

OUTCOME MEASURES:

1. Primary Outcome: Sleep Quality
Description: Measured by the Pittsburgh Sleep Quality Index (PSQI); Scores range from 0 to 21. Higher scores indicate poorer sleep quality. Scores >6 indicate poor sleep quality.
Time Frame: 4 months
Population: Individuals with outcome measured at 4 months.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | SleepTrackTXT2 | Text-Message Assessments Only
Number analyzed (Participants) | 16 | 27
score on a scale | 7.9 (3.6) | 6.5 (4.0)
Statistical Analysis 1: Comparison: SleepTrackTXT2 vs Text-Message Assessments Only; Test type: Superiority; p = 0.76, t-test, 2 sided; Two sample t-test on the change in sleep quality from baseline to 4 months

2. Secondary Outcome: Fatigue During Shiftwork
Description: Single item measure of fatigue taken at beginning, every 4-hours, and at the end of shifts. Scores range from 0 (Not at all) to 5 (Very much); higher scores indicate more fatigue.
Time Frame: Every 4 hours up to 12 hours within work shifts
Population: Participants with at least some intra-shift data on fatigue.
Measure: Least Squares Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | SleepTrackTXT2 | Text-Message Assessments Only
Number analyzed (Participants) | 35 | 41
score on a scale
  Start of Shift | 0.71 [0.36 to 1.06] | 0.79 [0.46 to 1.12]
  4 hours | 0.96 [0.61 to 1.31] | 1.10 [0.77 to 1.43]
  8 hours | 1.45 [1.10 to 1.80] | 1.79 [1.46 to 2.12]
  12 hours (end of shift) | 1.5 [1.14 to 1.84] | 2.19 [1.86 to 2.51]
Statistical Analysis 1: Comparison: SleepTrackTXT2 vs Text-Message Assessments Only; Test type: Superiority; p < 0.0001, Mixed Models Analysis — Test for group*time interaction

3. Secondary Outcome: Sleepiness During Shiftwork
Description: Single item measure of sleepiness taken at beginning, every 4-hours, and at the end of shifts. Scores range from 0 (Not at all) to 5 (Very much). Higher scores indicate more sleepiness.
Time Frame: Every 4 hours up to 12 hours within a work shift
Population: Individuals with shift data up to 30 days
Measure: Least Squares Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | SleepTrackTXT2 | Text-Message Assessments Only
Number analyzed (Participants) | 35 | 41
score on a scale
  Start of shift | 0.84 [0.49 to 1.19] | 0.82 [0.49 to 1.15]
  4 hours | 1.01 [0.66 to 1.35] | 1.29 [0.96 to 1.61]
  8 hours | 1.48 [1.12 to 1.83] | 2.01 [1.68 to 2.34]
  12 hours at shift end | 1.62 [1.27 to 1.97] | 2.50 [2.15 to 2.80]
Statistical Analysis 1: Comparison: SleepTrackTXT2 vs Text-Message Assessments Only; Test type: Superiority; p < 0.0001, Mixed Models Analysis; Test for group*time interaction

4. Secondary Outcome: Difficulty With Concentration During Shiftwork
Description: Single item measure of difficulty with concentration taken at beginning, every 4-hours, and at the end of shifts. Scores range from 0 (Not at all) to 5 (Very much). Higher scores indicate more difficulty with concentration.
Time Frame: Every 4 hours up to 12 hours at end of work shift
Population: Number with shift data at 30 days
Measure: Least Squares Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | SleepTrackTXT2 | Text-Message Assessments Only
Number analyzed (Participants) | 35 | 41
score on a scale
  Start of shift | 0.52 [0.19 to 0.86] | 0.46 [0.15 to 0.77]
  4 hours | 0.68 [0.35 to 1.02] | 0.71 [0.40 to 1.03]
  8 hours | 1.12 [0.78 to 1.45] | 1.27 [0.95 to 1.58]
  12 hours end of shift | 1.12 [0.79 to 1.46] | 1.76 [1.45 to 2.07]
Statistical Analysis 1: Comparison: SleepTrackTXT2 vs Text-Message Assessments Only; Test type: Superiority; p < 0.0001, Mixed Models Analysis; Test for group*time interaction

5. Secondary Outcome: Inter-Shift Recovery
Description: The Occupational Fatigue Exhaustion Recovery Scale Inter-shift Recovery Subscale. Scores range from 0 to 100. Scores 50-100 imply moderate to high recovery.
Time Frame: 4 months
Population: Participants with survey data at 4 months.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | SleepTrackTXT2 | Text-Message Assessments Only
Number analyzed (Participants) | 16 | 27
score on a scale | 51.7 (20.0) | 56.3 (18.8)
Statistical Analysis 1: Comparison: SleepTrackTXT2 vs Text-Message Assessments Only; Test type: Superiority; p = 0.91, t-test, 2 sided; Two sample t-test for change in Occupational Fatigue Exhaustion Recovery (OFER) inter-shift recovery between groups

ADVERSE EVENTS:
Time Frame: 4 months
Arm/Group | SleepTrackTXT2 | Text-Message Assessments Only
All-Cause Mortality (participants affected / at risk) | 0/39 | 0/44
Serious Adverse Events (participants affected / at risk) | 0/39 | 0/44
Other Adverse Events (participants affected / at risk) | 0/39 | 0/44

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-03-08): https://cdn.clinicaltrials.gov/large-docs/27/NCT02783027/Prot_SAP_000.pdf